CLINICAL TRIAL: NCT01795911
Title: A Phase 2B, Randomized Study to Evaluate the Safety and Efficacy of Pegylated Interferon Lambda (BMS-914143) Administered With Ribavirin Plus a Single Direct Antiviral Agent (BMS-790052 or BMS-650032) Versus Pegasys Administered With Ribavirin (Part A) and of Pegylated Interferon Lambda (BMS-914143) Administered With or Without Ribavirin Plus 2 Direct Antiviral Agents (BMS-790052 and BMS-650032) (Part B) in Chronic Hepatitis C Genotype-1 Treatment naïve Subjects
Brief Title: Safety Study of Pegylated Interferon Lambda Plus Single or 2 Direct Antiviral Agents With Ribavirin
Acronym: D-LITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI452-008 (Substudy Part C); 2010-022568-11 (EudraCT Number)
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; Ribavirin; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Substudy C: Pegylated Interferon Lambda+Ribasphere+Daclatasvir (Experimental): Pegylated Interferon Lambda 180 μg Solution, Subcutaneous Once weekly for 12 weeks;
  Ribasphere 1000 mg for subjects weighing < 75 kg and 1200 mg for subjects weighing ≥ 75 kg oral tablets per day [subjects should take either 400 mg for subjects < 75 kg or 600 mg ≥ 75 kg in the morning with food and 600 mg in the evening with food] for 12 weeks;
  Daclatasvir 60 mg oral tablet Once daily for 12 weeks
  Interventions: Biological: Pegylated Interferon Lambda; Drug: Ribasphere; Drug: Daclatasvir

INTERVENTIONS:
Biological: Pegylated Interferon Lambda
  Other Names: BMS-914143
Drug: Ribasphere
  Other Names: Ribavirin
Drug: Daclatasvir
  Other Names: BMS-790052

SUMMARY:
Substudy C: The purpose of this substudy is to determine whether Lambda combined with Ribavirin and Daclatasvir for 12 weeks is efficacious in treatment naïve subjects with genotype 1b chronic HCV infection

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C, Genotype 1
* HCV RNA >100,000 IU/mL at screening;
* Seronegative for Human immunodeficiency virus (HIV) and Hepatitis B surface antigen (HBsAg);
* Liver biopsy within prior 2 years; subjects with compensated cirrhosis can enroll and will be capped at approximately 10%

Exclusion Criteria:

* Any evidence of liver disease other than HCV;
* Co-infection with HIV;
* Diagnosed or suspected hepatocellular carcinoma;
* Medical history or laboratory value abnormalities that would prohibit the use of Pegylated Interferon Alpha-2a or Ribavirin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Antiviral activity, as determined by the proportion of non-cirrhotic HCV GT-1b subjects with 12-week sustained virologic response (SVR12), defined as HCV RNA < LLOQ target detected or not detected | Post-treatment Week 12
  HCV = Hepatitis C virus; GT = Geno Type; RNA = Ribonucleic acid; LLOQ = Lower limit of quantitation

SECONDARY OUTCOMES:
Proportion of non-cirrhotic HCV GT-1b subjects with eRVR, defined as HCV RNA < LLOQ target not detected | At Week 4 and Week 12
  eRVR = Extended rapid virologic response
Proportion of non-cirrhotic HCV GT-1b subjects with treatment-emergent cytopenic abnormalities (anemia as defined by Hb < 10 g/dL, and/or neutropenia as defined by ANC < 750 mm3, and/or thrombocytopenia as defined by platelets < 50,000 mm3) on treatment | On-treatment Weeks 1, 2, 4, 8, and 12
  Hb = Hemoglobin; ANC = Absolute neutrophil count
Proportion of non-cirrhotic HCV GT-1b subjects with on-treatment (maximum of 12 weeks) interferon-associated flu-like symptoms (pyrexia or chills or pain) | On-treatment Weeks 1, 2, 4, 8, and 12
Proportion of non-cirrhotic HCV GT-1b subjects with on-treatment (maximum of 12 weeks) interferon-associated musculoskeletal symptoms (arthralgia or myalgia or back pain) | On-treatment Weeks 1, 2, 4, 8, and 12
Proportion of non-cirrhotic HCV GT-1b subjects with SVR24, defined as HCV RNA < LLOQ target detected or not detected | Post-treatment follow-up Week 24
Frequency of deaths among non-cirrhotic HCV GT-1b subjects through the end of follow-up (maximum of 60 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12 and post-treatment weeks 4, 12, 24, 36 and 48
Frequency of Serious adverse events (SAEs) among non-cirrhotic HCV GT-1b subjects through the end of follow-up (maximum of 60 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12 and post-treatment weeks 4, 12, 24, 36 and 48
Frequency of drug related Adverse events (AEs) among non-cirrhotic HCV GT-1b subjects through the end of treatment (maximum of 12 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12
Frequency of dose reductions and discontinuations due to AEs among non-cirrhotic HCV GT-1b subjects through the end of treatment (maximum of 12 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12
Frequency of treatment emergent laboratory abnormalities among non-cirrhotic HCV GT-1b subjects through the end of treatment (maximum of 12 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12
Proportion of non-cirrhotic HCV GT-1b subjects with interferon-associated constitutional symptoms (fatigue or asthenia) through the end of treatment (maximum of 12 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12
Proportion of non-cirrhotic HCV GT-1b subjects with interferon-associated neurologic symptoms (headache or dizziness) through the end of treatment (maximum of 12 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12
Proportion of non-cirrhotic HCV GT-1b subjects with psychiatric symptoms (depression or irritability or insomnia) through the end of treatment (maximum of 12 weeks) | On-treatment Weeks 1, 2, 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Alamo Medical Research, San Antonio, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx